CLINICAL TRIAL: NCT04929418
Title: Differential Adaptation of Renal Function in Two Types of Intense Physical Exercise
Brief Title: Differential Adaptation of Renal Function in Intense Physical Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Collaborators: Gerencia Regional de Salud de Castilla y Leon (Other); Instituto de Investigación Biomédica de Salamanca (Other); Centro Regional de Medicina Deportiva de Castilla y León (Unknown)
Responsible Party: Principal Investigator, Armando Coca Rojo, MD, MSc, phD, Hospital Clínico Universitario de Valladolid
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PI-GR-18-914; GRS 1732A/18 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y León)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Trial participants will participate sequentially in two tests that involve high intensity physical exercise (10 km continuous running and 1.5 km continuous swimming). Both tests will be separated from each other a minimum of 30 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 km continuous running (Other): Participants will perform a test of 10 km coninuous running.
  Interventions: Other: 10 km continuous running; Other: 1.5 km continuous swimming
- 1.5 km swimming (Other): Participants will perform a test of 1.5 km coninuous swimming.
  Interventions: Other: 10 km continuous running; Other: 1.5 km continuous swimming

INTERVENTIONS:
Other: 10 km continuous running — Trial participants will perform a 10 km continuous running exercise
Other: 1.5 km continuous swimming — Trial participants will perform a 1.5 km continuous swimming exercise.

SUMMARY:
In recent years there has been a significant increase in the number of participants in high intensity and duration sports events. This type of physical exercise has been reported to lead to an apparently transitory deterioration in kidney function. The injury mechanisms involved in this process have not been fully studied, but several have been proposed as potential causes, such as tissue ischemia, disruption of the permeability of the glomerular basement membrane, damage to the ultra-structure of skeletal muscle, structural involvement of the renal parenchyma, exercise-associated hyperthermia or insufficient hydration during exercise.

Urinary biomarkers, which are a more precise tool than serum creatinine when it comes to detecting subclinical kidney damage, may be key to elucidate the characteristics of exercise-related kidney injury.

The aim of this study is to carry out an integrative analysis of the development of exercise-associated subclinical acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Able to understand the objectives of the study and to provide informed consent.
* Body mass index between 18.5 and 24.9 kg / m2
* Active sportsman/woman (defined as previous experience with the planned tests and performing vigorous-intensity aerobic activity at least three times per week).

Exclusion Criteria:

* History of chronic kidney disease, hypertension, uncontrolled diabetes (defined as fasting glucose levels ≥200 mg/dl or HbA1c ≥9%), peripheral vascular disease, heart disease, neurological disease or thyroid disease.
* Use of NSAIDs in the 72h prior to the test.
* Consumption of statins or anabolic steroids.
* Some kind of major physical injury in the four months prior to the tests.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Absolute change in urinary Neutrophil Gelatinase-Associated Lipocalin (NGAL) levels | 24 hours
Absolute change in urinary Kidney Injury Molecule-1 (KIM-1) levels | 24 hours

SECONDARY OUTCOMES:
Absolute change in serum creatinine levels | 24 hours
Absolute change in proteinuria | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No